CLINICAL TRIAL: NCT03903003
Title: In the Study; Preoperative Highflow Nasal Oxygen Application in Cesarean Under General Anesthesia and Its Effects on Newborn.
Brief Title: Preoperative Highflow Nasal Oxygen Application in Cesarean Under General Anesthesia and Its Effects on Newborn.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, EMİNE YURT, clinical researcher, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: KIA 2018/506
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Cesarean Delivery Affecting Newborn
Keywords: high flow nasal oxygen (POİNT)
MeSH Terms: interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoxygenation mask applied to the cesarean (Active Comparator): In order to protect the mother from hypoxia, preoxygenation is performed with face mask before induction of anesthesia.
  Interventions: Device: Face mask
- high flow nasal oxygenation applied to the ceserian (Active Comparator): In order to protect the mother from hypoxia, preoxygenation is performed with high flow nasal oxygenation mask before induction of anesthesia.
  Interventions: Device: high flow nasal oxygen device (POİNT)

INTERVENTIONS:
Device: high flow nasal oxygen device (POİNT) — With POINT device (peri-operative insufflatory nasal therapy); patients are heated at higher flow and applied to humidified oxygen.
  Arms: high flow nasal oxygenation applied to the ceserian
Device: Face mask — In order to protect the mother from hypoxia, preoxygenation is performed with face mask before induction of anesthesia.
  Arms: preoxygenation mask applied to the cesarean

SUMMARY:
Preoperative Highflow Nasal Oxygen Application in Cesarean Under General Anesthesia and Its Effects on Newborn.

DETAILED DESCRIPTION:
Patients who will undergo caesarean section under general anesthesia will be included in the study.

In the study; preoxygenation is applied to the caesarean sections under general anesthesia in two ways. Group1 includes preoxygenation masked patients.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old;
* Patients undergoing elective ceserian operation

Exclusion Criteria:

* Patients who refuse to participate in the study;
* Patients under emergency conditions.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
durations of stay | 24 hours
  compare the durations of stay in the intensive care unit and in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yılmaz, Study Director — HEALTH AND SCİENCE UNIVERSITY MEDICAL SCHOOL
Locations (1):
- Kocaeli Derince Education and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided